CLINICAL TRIAL: NCT03047213
Title: An Open Label, Multicenter, Single Arm Phase II Study to Evaluate the Activity and Tolerability of the Novel mTOR Inhibitor, MLN0128 (TAK-228), in Patients With Locally Advanced or Metastatic Transitional Cell Carcinoma of the Urothelial Tract Whose Tumors Harbor a TSC1 and/or a TSC2 Mutation
Brief Title: Sapanisertib in Treating Patients With Locally Advanced or Metastatic Bladder Cancer With TSC1 and/or TSC2 Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00121; NCI-2015-00121 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1505015958; 2000021268; 9767 (Other: Yale University Cancer Center LAO); 9767 (Other: CTEP); UM1CA186689 (NIH); NCT03108261 (obsolete NCT alias)
Record Dates: First submitted 2017-02-07; First posted 2017-02-08 (Estimated); Results first posted 2025-02-11 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Bladder Urothelial Carcinoma; Metastatic Transitional Cell Carcinoma; Metastatic Urothelial Carcinoma; Recurrent Bladder Carcinoma; Stage III Bladder Urothelial Carcinoma AJCC v6 and v7; Stage IV Bladder Urothelial Carcinoma AJCC v7
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sapanisertib) (Experimental): Patients receive sapanisertib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sapanisertib

INTERVENTIONS:
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228

SUMMARY:
This pilot phase II trial studies how well sapanisertib works in treating patients with bladder cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or other places in the body (metastatic) with tuberous sclerosis (TSC)1 and/or TSC2 mutations (changes in deoxyribonucleic acid [DNA]). Sapanisertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) defined as complete response (CR) and partial response (PR) in patients with locally advanced or metastatic transitional cell carcinoma (TCC) harboring a TSC1 mutation.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of sapanisertib (MLN0128) (TAK-228) in patients with locally advanced or metastatic TCC harboring a TSC1 or TSC2 mutation.

II. To evaluate progression free survival (PFS) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To determine the ORR in patients with locally advanced or metastatic TCC harboring a TSC2 mutation.

II. To evaluate toxicity, PFS, and OS in TSC2 mutation patients.

OUTLINE:

Patients receive sapanisertib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Must have a histologically confirmed transitional cell carcinoma (TCC, also known as urothelial carcinoma), locally advanced or metastatic
* Patient must have TCCs tumors harboring a TSC1 or TSC2 mutation identified by a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory
* Unless the pre-screening was performed at Yale Clinical Molecular Pathology Lab (YCMPL), patients must have TCC tumor tissue available for submission in a form of at least 10 unstained slides or formalin-fixed paraffin-embedded (FFPE) block (FFPE block highly recommended and preferred) along with a buccal swab; if the number of slides is less than 10, a biopsy should be considered; if a biopsy is deemed unsafe, the case may be discussed with the study principal investigator (PI) and approval must be given for eligibility
* Patient must have developed disease progression during or following treatment with at least one platinum-containing regimen (e.g., gemcitabine/cisplatin [GC], methotrexate-vinblastine-doxorubicin-cisplatin [MVAC], carboplatin, gemcitabine [CarboGem]) for inoperable locally advanced or metastatic urothelial carcinoma or disease recurrence, or must be unfit or ineligible for cisplatin-based chemotherapy; there is no restriction on the number of prior lines of chemotherapeutics agents received

  * Patients who progressed within 12 months of treatment with a platinum-containing neoadjuvant or adjuvant regimen are considered second-line patients; therefore, these patients may be also eligible
  * Patients who are unfit or ineligible for cisplatin-based chemotherapy as defined by any one of the following criteria are eligible for this trial:

    * Eastern Cooperative Oncology Group (ECOG) performance score of 2
    * Creatinine clearance < 60 mL/min
    * A hearing loss (measured by audiometry) of 25 dB at two contiguous frequencies
    * Grade >= 2 peripheral neuropathy
* ECOG performance status =< 2 (Karnofsky >= 60 %)
* Life expectancy of greater than 12 weeks
* Hemoglobin >= 9 g/dL
* Fasting serum glucose =< 130 mg/dL
* Glycosylated hemoglobin measurement (HbA1c) < 7.0%
* Fasting triglycerides =< 300 mg/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN) and =< 5 ULN if liver metastases are present
* Creatinine =< 1.5 x upper normal institutional limits (UNL) OR creatinine clearance >= 40 mL/min based either on Cockcroft-Gault estimate or based on urine collection (12 or 24 hour)
* Patients with controlled diabetes are allowed on study; controlled diabetes is defined as fasting blood sugar (FBS) = 130 mg/dL or less, and patients whose FBS can be brought in this range with medical therapy are eligible for trial inclusion
* The effects of MLN0128 (TAK-228) on the developing human fetus are unknown; fertility and developmental studies with MLN0128 (TAK-228) have not been conducted; on the basis of potential hazard of other mTOR inhibitors (i.e., rapamycin and other rapalogs) on the developing fetus, women of childbearing age should avoid becoming pregnant while taking any mTOR inhibitor including MLN0128 (TAK-228)

  * Female patients must:

    * Be postmenopausal for at least 1 year before the screening visit, OR
    * Be surgically sterile, OR
    * If they are of childbearing potential, agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer, as mandated by local labeling [e.g., United States product insert [USPI], summary of product characteristics [SmPC], etc.;]) after the last dose of study drug, OR
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient; NOTE: periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception; female and male condoms should not be used together
  * Male patients, even if surgically sterilized (i.e., status postvasectomy), must:

    * Agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient (NOTE: periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception; female and male condoms should not be used together)
    * AND agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug
* Ability to swallow oral medications
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, immunotherapy, or investigational therapy, within 4 weeks (6 weeks for nitrosoureas or mitomycin C), or palliative radiotherapy within 2 weeks prior to the first dose of the study drug
* Patients who have not recovered from adverse events due to prior anti-cancer therapy to grade 1 or baseline; patients with stable, controlled grade 2 adverse events (AEs) such as peripheral neuropathy, hypothyroidism, hypertension, adrenal insufficiency or alopecia are allowed after discussing with the PI
* Patients with known symptomatic, untreated central nervous system (including brain, spinal cord); patients who have a history of brain/central nervous system (CNS) metastasis are eligible for the study provided that all the following criteria are met:

  * Brain/CNS metastases which have been treated
  * No evidence of disease progression for >= 3 months before the first dose of study drug
  * No hemorrhage after treatment
  * Off-treatment with dexamethasone for 4 weeks before administration of the first dose of TAK-228
  * No ongoing requirement for dexamethasone or anti-epileptic drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN0128 (TAK-228)
* Subjects who are on systemic corticosteroids (intravenous (IV) or oral steroids, excluding inhaled, topical or ophthalmic corticosteroids), or anti-epileptic drugs for treated brain metastasis
* Subjects taking strong inhibitors and/or inducers of cytochrome P450 (CYP) 3A4, CYP2C19 or CYP2C9 within 1 week preceding the first dose of MLN0128 (TAK-228); if a subject requires treatment with strong inhibitors and/or inducers of CYP3A4, CYP2C19 and/or CYP2C9, alternative treatment must be considered; if no alternative is available, one such medication may be allowed after discussing with the study principle investigator
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding rate controlled atrial fibrillation/flutter), or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded from this study because fertility and developmental studies with MLN0128 (TAK-228) have not been conducted and there is a potential risk for adverse events including teratogenicity and risk of abortion; breastfeeding should be discontinued if the mother is treated with MLN0128 (TAK-228)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MLN0128 (TAK-228); however, HIV patients treated with regimens that have low CYP450 inhibition may be allowed as long as the patient's general health and CD4 counts are within acceptable levels
* Patients with baseline prolongation of the rate-corrected QT interval (QTc) (e.g., repeated demonstration of QTc interval > 480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes)
* Patients with untreated or active hepatitis B or C infection
* Significant active cardiovascular or pulmonary disease at the time of study entry, including

  * Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg)
  * Pulmonary hypertension
  * Uncontrolled asthma or oxygen (O2) saturation < 90% by ABG (arterial blood gas) analysis or pulse oximetry on room air
  * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement
  * Medically significant (symptomatic) bradycardia
* Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of MLN0128 (TAK-228)
* Concomitant administration of any proton pump inhibitor (PPI) is not permitted during the study; patients receiving PPI therapy before enrollment must stop using the PPI for 7 days before their first dose of study drugs
* History of any of the following within the last 6 months prior to study entry:

  * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
  * Ischemic cerebrovascular event, including transient ischemic attack (TIA) and artery revascularization procedures
  * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
  * Pulmonary embolism
  * New York Heart Association (NYHA) class III or IV heart failure
  * Placement of a pacemaker for control of rhythm
* Subjects who have initiated treatment with bisphosphonates less than 30 days prior to the first administration of MLN0128 (TAK-228); concurrent bisphosphonate use is only allowed if the bisphosphonate was initiated at least 30 days prior to the first administration of MLN0128 (TAK-228)
* Patients who received prior PI3K, AKT or mTOR inhibitors are not allowed
* Patients who received radiation therapy within the last 4 weeks; radiation exposure may not exceed 30% of marrow area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2026-11-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Kim, Principal Investigator — Yale University Cancer Center LAO
Locations (20):
- United States (20):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Sapanisertib): TSC Mutation 1; TSC Mutation 2: Patients receive sapanisertib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Sapanisertib: Given PO
Period: Overall Study
Arm/Group | Treatment (Sapanisertib): TSC Mutation 1 | TSC Mutation 2
Started | 14 | 3
Completed | 10 | 3
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Sapanisertib): TSC Mutation 1 | TSC Mutation 2 | Total
Number analyzed (Participants) | 14 | 3 | 17
Age, Continuous [Median (Full Range); unit: years] | 68.5 [53 to 84] | 61 [55 to 78] | 67 [53 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 13 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 3 | 15
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 3 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 3 | 17
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG Performance Status Scale ranges from 0 to 5, with lower scores indicating better functional status.
  0:Fully active, able to carry on all pre-disease activities without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out light work.
  2. Ambulatory and capable of self-care but unable to carry out work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care. Confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry out any self-care. Totally confined to bed or chair.
  5. Dead.
  Participants
    0 | 5 | 1 | 6
    1 | 7 | 2 | 9
    2 | 2 | 0 | 2
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (TSC1 Patients)
Description: Overall Response Rate is the proportion of the patients with either complete response (CR) or partial response (PR) by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) version 1.1. Complete Response (CR) is defined as disappearance of all target lesions and partial response (PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Overall Response Rate is the proportion of the patients with either complete response (CR) or partial response (PR) by Response Evaluation Criteria. In Solid Tumors Criteria (RECIST) version 1.1. Complete Response (CR) is defined as disappearance of all target lesions and partial response (PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 4 weeks after last dose of study treatment (approximately 19 weeks)
Population: 12 of 14 patients were evaluable for the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sapanisertib): TSC Mutation 1
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Incidence of Toxicity (TSC1 Patients)
Description: Presented are the most frequently occurring adverse events (25% of patients or greater)
Time Frame: Up to 4 weeks after last dose of study treatment (approximately 19 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sapanisertib): TSC Mutation 1
Number analyzed (Participants) | 12
Participants
  Hyperglycemia | 11
  Creatinine increased | 7
  Hypoalbuminemia | 7
  Anemia | 6
  AST increased | 5
  diarrhea | 5
  lymphocyte count decreased | 5
  rash | 5
  Alkaline phosphatase increased | 4
  Abdominal pain | 3
  Anorexia | 3
  Fatigue | 3
  Hyperkalemia | 3
  hypomagnesemia | 3
  Hypophosphatemia | 3
  nausea | 3
  platelet count decreased | 3
  urinary tract infection | 3
  vomiting | 3
  weight loss | 3

3. Secondary Outcome: Progression-free Survival (PFS) (TSC1 Patients)
Description: The censored PFS distributions will each be estimated by the Kaplan-Meier (K-M) survivorship function. Point estimates and 90% (2-sided) CIs will be computed for all estimable summary statistics, e.g., the median, 6-month rate, 12-month rate, etc. Upon results entry, no patients had reached 6 or 12 months PFS and the outcome and timeframe have been updated. Progression-free survival (PFS) is defined as the duration of time from start of treatment to date of progression or death, whichever occurs first. Progression by RECIST v1.1 criteria is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Time from start of treatment to date of progression or death- (approximately 19 weeks)
Population: 12 of 14 patients were evaluable
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Sapanisertib): TSC Mutation 1
Number analyzed (Participants) | 12
days | 54 [10 to 127]

4. Secondary Outcome: Overall Survival (OS) (TSC1 Patients)
Description: The censored OS distributions will each be estimated by the K-M survivorship function. Point estimates and 90% (2-sided) CIs will be computed for all estimable summary statistics, e.g., the median, 6-month rate, 12-month rate, etc.
Time Frame: Time from start of treatment to time of death from any cause, up to approximately 9 months
Population: 12 of 14 patients were evaluable
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Sapanisertib): TSC Mutation 1
Number analyzed (Participants) | 12
days | 114 [32 to 192]

5. Other Pre Specified Outcome: Overall Response Rate (TSC2 Patients)
Time Frame: Up to 4 weeks after last dose of study treatment (approximately 19 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | TSC Mutation 2
Number analyzed (Participants) | 3
Participants | 0

6. Other Pre Specified Outcome: Incidence of Toxicity (TSC2 Patients)
Description: The occurrence rate of each specific type of toxicity at a certain severity grade will be described by point estimates and Wilson type 90% (2-sided) CIs.
Time Frame: Up to 4 weeks after last dose of study treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Progression-free Survival (TSC2 Patients)
Description: The censored PFS distributions will each be estimated by the K-M survivorship function. Point estimates and 90% (2-sided) CIs will be computed for all estimable summary statistics, e.g., the median, 6-month rate, 12-month rate, etc.
Time Frame: Time from start of treatment to date of progression or death, whichever occurs first, assessed up to 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Overall Survival (TSC2 Patients)
Description: as for outcome 4
Time Frame: Time from start of treatment to time of death from any cause, assessed up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 9 months
Arm/Group | Treatment (Sapanisertib): TSC Mutation 1 | TSC Mutation 2
All-Cause Mortality (participants affected / at risk) | 10/12 | 3/3
Serious Adverse Events (participants affected / at risk) | 6/12 | 2/3
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sapanisertib): TSC Mutation 1 (N=12) | TSC Mutation 2 (N=3)
Creatinine increased (Renal and urinary disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
platelet count decreased (Blood and lymphatic system disorders) | 1 | 0
AKI (Renal and urinary disorders) | 2 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
dehydration (Metabolism and nutrition disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 1 | 0
bowel obstruction (Gastrointestinal disorders) | 1 | 0
GI hemorrhage (Gastrointestinal disorders) | 1 | 0
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
syncope (Nervous system disorders) | 1 | 0
urinary tract obstruction (Renal and urinary disorders) | 1 | 0
ALT increased (Hepatobiliary disorders) | 0 | 1
AST increase (Hepatobiliary disorders) | 0 | 1
urinary tract injection (Infections and infestations) | 0 | 2
Alkaline phosphatase increased (Hepatobiliary disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sapanisertib): TSC Mutation 1 (N=12) | TSC Mutation 2 (N=3)
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Activated PTT prolonged (Investigations) | 1 | 0
AKI (Renal and urinary disorders) | 2 | 0
Alkaline phosphatase increased (Hepatobiliary disorders) | 4 | 1
ALT increased (Hepatobiliary disorders) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 6 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
AST increased (Hepatobiliary disorders) | 5 | 2
back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Blood bilirubin increased (Hepatobiliary disorders) | 1 | 2
bowel obstruction (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Cholesterol high (Metabolism and nutrition disorders) | 2 | 0
constipation (Gastrointestinal disorders) | 1 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Creatinine increased (Renal and urinary disorders) | 7 | 1
dehydration (Metabolism and nutrition disorders) | 2 | 0
diarrhea (Gastrointestinal disorders) | 5 | 0
Dizziness (Nervous system disorders) | 2 | 0
drop foot (Nervous system disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
edema (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fatigue (General disorders) | 3 | 1
fever (Infections and infestations) | 0 | 1
Flank pain (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
GI hemorrhage (Gastrointestinal disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
hypotension (Vascular disorders) | 1 | 0
INR increased (Investigations) | 0 | 1
insomnia (Psychiatric disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
lipase increase (Investigations) | 1 | 0
lymphocyte count decreased (Blood and lymphatic system disorders) | 5 | 0
malaise (General disorders) | 2 | 0
mucositis oral (Gastrointestinal disorders) | 2 | 0
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
nausea (General disorders) | 3 | 0
non-cardiac chest pain (General disorders) | 1 | 0
pain (General disorders) | 2 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
platelet count decreased (Blood and lymphatic system disorders) | 3 | 0
proteinuria (Renal and urinary disorders) | 1 | 0
pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
rash (Skin and subcutaneous tissue disorders) | 5 | 0
sepsis (Infections and infestations) | 0 | 1
sinus bradycardia (Cardiac disorders) | 1 | 0
syncope (Nervous system disorders) | 1 | 0
urinary tract infection (Infections and infestations) | 3 | 2
urinary tract obstruction (Renal and urinary disorders) | 1 | 0
vomiting (General disorders) | 3 | 0
weight loss (Metabolism and nutrition disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03047213/Prot_SAP_000.pdf